CLINICAL TRIAL: NCT03488355
Title: Modified Reporting of Positive Urine Cultures Collected From Indwelling Catheters, a Randomized Controlled Trial
Brief Title: Modified Reporting From Indwelling Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Peter Daley, Associate Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUN-3
Record Dates: First submitted 2018-03-26; First posted 2018-04-05 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-04

CONDITIONS: Urinary Tract Infections
Keywords: Catheter
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Reporting (Experimental): Modified laboratory report
  Interventions: Other: Modified laboratory report
- Standard Reporting (No Intervention): Standard laboratory report

INTERVENTIONS:
Other: Modified laboratory report — Report from microbiology laboratory: "This POSITIVE urine culture collected from an indwelling catheter may represent asymptomatic bacteriuria or urinary tract infection. If urinary tract infection is suspected clinically, please call the microbiology laboratory for identification and susceptibility results."
  Arms: Modified Reporting

SUMMARY:
Positive urine cultures collected from indwelling catheters from inpatients will be randomized to standard reporting or modified reporting. Physician antibiotic treatment decisions will be prospectively observed and determined to be appropriate or inappropriate. The hypothesis is that modified reporting will lead to an increase in the percentage of appropriate therapy without an increase in pyelonephritis or sepsis.

DETAILED DESCRIPTION:
The proposed study is a randomized trial of two methods of laboratory reporting in which physicians are the main research participants. At the time of positive urine culture results, the patient will be randomized by computer generated random number placed into serially numbered sealed, opaque envelopes into two equal groups. One group will receive modified reporting, with a report that states "This POSITIVE urine culture collected from an indwelling catheter may represent asymptomatic bacteriuria or urinary tract infection. If urinary tract infection is suspected clinically, please call the microbiology laboratory for identification and susceptibility results." The other group will receive conventional reporting of identification and susceptibility. Physicians will then have the option of calling the laboratory to receive the results or not. Complete results will be released by telephone and laboratory information system to physicians who call to request them. Physicians will be informed about the study prior to initiation, and debriefed about the study after the results have been collected.

Inclusion criteria will include consecutive positive urine cultures collected from indwelling catheters among patients admitted to acute care, that are greater than or equal to 18 years of age. Inpatients must be admitted to Health Sciences Center or St. Clare's Mercy hospitals only, in order to facilitate access to inpatient records.

Exclusion criteria will include pregnancy, antibiotic treatment at the time of collection, patients in the Intensive Care Unit and patients with blood neutrophils <1.0 within 7 days, which will help protect immunocompromised individuals.

Investigators will review patient charts at 24 and 72 hours and 7 days after collection. After randomization and reporting, a physician investigator will assess inpatients for the true diagnosis of asymptomatic bacteriuria (AB) or urinary tract infection (UTI). Health records will be accessed including demographics, treatment decisions and outcomes (untreated UTI or pyelonephritis). Frequency of physician calls requesting complete reporting will be recorded.

The research hypothesis is that restricted reporting will reduce the rate of inappropriate treatment prescribed by physicians. Among inpatients, the expected rate of inappropriate treatment in the control group will be 50 percent, and 20 percent in the intervention group. Accepting a risk of type 1 error of five percent, and a risk of type 2 error of twenty percent, the study will recruit 72 patients. In order to account for missing data, recruitment will be increased to 100 patients. The statistical test to be used is a comparison of proportions between two groups (T test, two sided analysis). An intention to treat analysis including all patients randomized will be performed.

Physicians must remain unaware of the research project so that their treatment decisions are unbiased. However, a general notice will be sent to all physicians regarding the study design, and a debrief will be provided in which study results are presented and the option to withdraw data will be provided. This will cause physicians to feel less deceived while still not informing them of the study and thus will not change their behavior.

Physicians of discharged inpatients will be contacted at 7 days to assess for adverse events. Because recruitment will be brief, it is unlikely that physicians will have a second patient in the study.

Ethics permission will be sought from the local ethics board. Consent of patients or physicians will not be requested. In compliance with ethics requirements, participants will experience no more than minimal risk. If an adverse event occurs, the patient will be removed from the study immediately and given standard treatment. Physician consent will not be requested, as awareness of the study would bias treatment decisions.

The benefit of this study to patients includes a reduction in adverse events caused by inappropriate treatment. The risk to patients includes possible untreated UTI. The benefit to physicians includes education toward appropriate treatment of AB. The risk to physicians includes additional effort to access laboratory results for UTI.

Data collection will use a paper case report form, and entry into a password protected online database. Analysis will be performed using SPSS 20.0 (IBM). The only expense of the project will be the graduate student to collect the data, perform the analysis and write the manuscript. The manuscript will be published in a peer-reviewed journal and presented at a national conference.

ELIGIBILITY:
Inclusion Criteria:

* consecutive positive urine cultures collected from indwelling catheters in inpatients that are greater than or equal to 18 years of age.
* admitted to Health Sciences Center or St. Clare's Mercy hospitals only

Exclusion Criteria:

* pregnancy
* antibiotic treatment at the time of collection
* patients in the Intensive Care Unit
* blood neutrophils count <1.0 x 10E9/l, within 7 days of urine collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Barrett, MD, Principal Investigator — Memorial University
Locations (1):
- Health Sciences Center, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pratt CL, Rehan Z, Xing L, Gilbert L, Fillier B, Barrett B, Daley P. Modified reporting of positive urine cultures to reduce inappropriate antibiotic treatment of catheter-associated asymptomatic bacteriuria (CA-ASB) among inpatients, a randomized controlled trial. Infect Control Hosp Epidemiol. 2021 Oct;42(10):1221-1227. doi: 10.1017/ice.2020.1397. Epub 2021 Jun 4. PMID 34085614

RESULTS

PARTICIPANT FLOW:
Groups:
- Modified Reporting: Modified laboratory report
  Modified laboratory report: Report from microbiology laboratory: "This POSITIVE urine culture collected from an indwelling catheter may represent asymptomatic bacteriuria or urinary tract infection. If urinary tract infection is suspected clinically, please call the microbiology laboratory for identification and susceptibility results."
  This intervention is not a drug or device, but a method of reporting of a laboratory report.
Period: Overall Study
Arm/Group | Modified Reporting | Standard Reporting
Started | 54 | 46
Completed | 54 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Reporting | Standard Reporting | Total
Number analyzed (Participants) | 54 | 46 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (12.6) | 73.3 (13.7) | 72.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 18 | 46
  Male | 26 | 28 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 54 | 46 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Appropriate Treatment
Description: Untreated catheter-associated asymptomatic bacteriurias, plus treated catheter-associated urinary tract infections, divided by total patients.
Time Frame: 7 days after positive urine culture
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Reporting | Standard Reporting
Number analyzed (Participants) | 54 | 46
Participants | 31 | 23
Statistical Analysis 1: Comparison: Modified Reporting vs Standard Reporting; Test type: Superiority; p = 0.45, t-test, 2 sided; Risk Ratio (RR) = 1.15

2. Secondary Outcome: Death
Description: All-cause mortality
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Reporting | Standard Reporting
Number analyzed (Participants) | 54 | 46
Participants | 4 | 3

3. Secondary Outcome: Adverse Events
Description: Number of participants with adverse events.
Time Frame: 7 days after positive urine culture
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Reporting | Standard Reporting
Number analyzed (Participants) | 54 | 46
Participants | 13 | 19

ADVERSE EVENTS:
Time Frame: Seven days
Description: Number of patients with adverse event
Arm/Group | Modified Reporting | Standard Reporting
All-Cause Mortality (participants affected / at risk) | 4/54 | 3/46
Serious Adverse Events (participants affected / at risk) | 3/54 | 0/46
Other Adverse Events (participants affected / at risk) | 13/54 | 19/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Reporting (N=54) | Standard Reporting (N=46)
Bacteremia (Infections and infestations) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Reporting (N=54) | Standard Reporting (N=46)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Auditory Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Candidemia (Infections and infestations) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Decreased level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Decreased white blood cell count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Edema (General disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Fluid Overload (General disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypokalemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Increased liver enzymes (General disorders) | 0 (0) | 1 (1)
Penis discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory secretions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin tear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shortness of breath (General disorders) | 1 (1) | 1 (1)
Suicidality (Psychiatric disorders) | 1 (1) | 0 (0)
Suprapubic tenderness (General disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/55/NCT03488355/Prot_SAP_000.pdf